CLINICAL TRIAL: NCT00594048
Title: The Effects of Device-guided Breathing Exercises on Blood Pressure in Patients With Hypertension. A Randomized, Single-blind, Controlled Trial
Brief Title: The Effects of Device-guided Breathing Exercises on Blood Pressure in Patients With Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical Research Foundation, The Netherlands (Other)
Responsible Party: Prof. dr. H.J.G. Bilo, Diabetes Centre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 07.1069; NL20147.075.07
Record Dates: First submitted 2008-01-04; First posted 2008-01-15 (Estimated); Last update posted 2011-10-26 (Estimated); Status verified 2011-10

CONDITIONS: Hypertension
Keywords: high blood pressure
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): 15 hypertensive patients use the Resperate for 9 weeks and measure their blood pressure before and after using this device
  Interventions: Device: Resperate
- 2 (Active Comparator): 15 patients use a discman with freely chosen music for 9 weeks and measure their blood pressure before and after use of this device
  Interventions: Device: discman with freely chosen music

INTERVENTIONS:
Device: Resperate — Use of the device 15 minutes a day for 9 weeks
  Other Names: device-guided breathing
  Arms: 1
Device: discman with freely chosen music — Use the discman 15 minutes a day for 9 weeks
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether breathing-exercises with the Resperate or listening to a discman with freely chosen music are effective in the treatment of hypertension

DETAILED DESCRIPTION:
Hypertension is an important risk factor for the development of macrovascular events. Lowering blood pressure leads to a reduced risk of developing these complications. To treat hypertension effectively you can use blood pressure lowering drugs, but it is also important to use proven and safe non-pharmacological interventions. It is suggested that Breathing Rate and Systolic Blood Pressure can be linked directly together by the baroreflex. With the use of the Resperate, people will lower their breathing rate by breathing similar to music patterns which could theoretically lead, through the described link, to blood pressure reduction. Patients will be randomize into two groups: one will get a discman with freely chosen music and the other the Resperate. Patients are instructed to use the breathing device or discman for 15 minutes at about the same time every day during the 9 week study period, except for the first week.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old
* Known hypertension with a SBP between 130-170 mmHg at previous visit to the internal outpatient department and at the last visit to the internist
* Treated with one or more anti-hypertensive drugs, which have not been changed for the preceding three months
* At Baseline the SBP should be between 140-160 mmHg

Exclusion Criteria:

* Patients with known diabetes
* Patients with heart failure (NYHA III-IV)
* Patients with pulmonary disease
* Patients with insufficient knowledge of the Dutch language to understand the requirements of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2008-01; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Systolic Blood Pressure | 9 weeks

SECONDARY OUTCOMES:
Quality of life | 9 weeks
Diastolic Blood Pressure | 9 weeks

CONTACTS AND LOCATIONS:
Overall Officials: N. Kleefstra, MD, Principal Investigator — Diabetes Centre, Isala Clinics, Zwolle; S.J.J. Logtenberg, MD, Principal Investigator — Diabetes Centre, Isala Clinics, Zwolle; K.H. Groenier, PhD, Principal Investigator — University of General Practice, UMCG Groningen; S.T. Houweling, MD PhD, Principal Investigator — Langerhans Medical Research Group; H.J.G. Bilo, MD PhD RFCP, Study Chair — Diabetes Centre, Isala Clinics, Zwolle
Locations (1):
- Diabetes Centre Zwolle, Zwolle, Overijssel, Netherlands

REFERENCES:
- [Derived] Altena MR, Kleefstra N, Logtenberg SJ, Groenier KH, Houweling ST, Bilo HJ. Effect of device-guided breathing exercises on blood pressure in patients with hypertension: a randomized controlled trial. Blood Press. 2009;18(5):273-9. doi: 10.3109/08037050903272925. PMID 19919399